CLINICAL TRIAL: NCT05235802
Title: Long-term Follow-up in Severe Traumatic Brain Injury
Acronym: LONG-TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eric Thelin, Principal Investigator (MD, PhD), Associate Professor, Karolinska University Hospital
Other Study IDs: 2021-02010; 4-1857 /2021 (Other: Karolinska Institutet); K 2021-5631 (Other: Karolinska University Hospital)
Record Dates: First submitted 2021-08-24; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury; Neurodegenerative Diseases; Chronic Traumatic Encephalopathy
Keywords: Fluid biomarkers; Neuroinflammatory process; Auto-immunity; Structural imaging; Clinical assessment; Long-term follow-up
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurodegenerative Diseases; Chronic Traumatic Encephalopathy | interventions — Magnetic Resonance Imaging; Blood Specimen Collection; Cerebrospinal Fluid Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, blood (whole blood, serum and plasma).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with traumatic brain injury about 10 years ago: Patients that had suffered a TBI and being managed at the Neurosurgical Department at the Karolinska University Hospital between 2007 and 2015.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI) (including functional MRI); Diagnostic Test: Blood sampling (serum/plasma preparation); Diagnostic Test: Cerebrospinal fluid (CSF); Diagnostic Test: Clinical assessments / questionnaires

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) (including functional MRI) — Patients will undergo magnetic resonance imaging including the following protocols:
  * 3D T1w MPRAGE
  * 3D T2w FLAIR SPACE
  * 3D T2w SPACE
  * 3D T1w PSIR (cortical visualization)
  * 2D synthetic MRI (quantitative T1, T2, PD and myelin quantification)
  * Resting-state fMRI (6 min, human connectome protocol, 2 mm iso)
  * 3D SWI
  * DWI b1000 32 directions and b3000 64 directions.
Diagnostic Test: Blood sampling (serum/plasma preparation) — Blood will be screened for genetic modifications. Serum will be analyzed for auto-antibodies and other inflammatory and neurodegenerative biomarkers.
Diagnostic Test: Cerebrospinal fluid (CSF) — CSF will be analyzed for inflammatory and neurodegenerative biomarkers.
Diagnostic Test: Clinical assessments / questionnaires — * Glasgow Outcome Scale Extended (functional outcome)
  * Short-Form 36 (quality of life),
  * EQ-5D (quality of life),
  * Mini-Mental State Extended (MMSE) (mental state assessment).
  * Barthel Index (daily living disabilities),
  * Montgomery-Åsberg Depression Score (MADRS-S) (level of depression)
  * Fatigue Severity Scale (FSS) (level of fatigue)
  Other than that, neurological assessments focusing on the Unified Parkinson's Disease Rating Scale (UPDRS) will be performed.

SUMMARY:
The underlying pathophysiology following traumatic brain injury (TBI) in how different neurodegenerative conditions are developed are still unknown. Different neuroinflammatory and neurodegenerative pathways have been suggested.

The goal of this study is to follow-up patients that have been treated for TBI at the neurosurgical department about 10-15 years after their initial injury, in order to analyze fluid biomarkers of inflammation, injury and degeneration and associate these with structural imaging and long-term functional outcome.

The investigators aim to invite about 100 patients back and perform advanced magnetic resonance imaging protocols, sample cerebrospinal fluid and blood for different bio- and inflammatory markers, study genetic modifications and associate it with outcomes being assessed through questionnaires.

The investigators' hypothesis is that patients with ongoing inflammatory processes will present with more fluid biomarkers of neurodegeneration, worse clinical presentation and also more structural/atrophic signs on imaging. This will result in an increased understanding of the interplay between neuroinflammation and neurodegeneration in chronic TBI, as well as a panel of tentative biomarkers that could be used to assess level of disability following TBI and chronic traumatic encephalopathy (CTE).

ELIGIBILITY:
Inclusion Criteria:

* Having suffered a traumatic brain injury and being treated at the Karolinska University Hospital between 2007 and 2015.
* Age >18 years of age

Exclusion Criteria:

- Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that had suffered a traumatic brain injury and registered at our local trauma database will be sent a letter asking them for participation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
GOSE vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Glasgow Outcome Score extended (1-8) will be associated alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (affected voxels).
Barthel Index vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Barthel Index (0-100) will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (affected voxels).
Fatigue Severity Scale vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Fatigue Severity Scale (9-63) will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (affected voxels).
MOCA vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Montreal Cognitive Assessment (MoCA) will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (MOCA score vs affected voxels).
SF-36 vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Short-Form 36 will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (SF-36 score vs affected voxels on MRI).
EQ-5D vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Health-related quality of life (EQ-5D) will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (EQ5D score vs affected voxels on MRI).
MADRS vs structural outcome | Assessed at the chronic time-point (10-15 years after injury).
  Montgomery-Åsberg depression rating scale (MADRS) will be associated with alterations at axonal and myelin integrity as assessed by magnetic resonance imaging (MADRS score vs affected voxels).
Structural outcome vs proteomic markers in serum | Assessed at the chronic time-point (10-15 years after injury).
  Alterations at axonal and myelin integrity as assessed by magnetic resonance imaging will be associated with a proteomic profiling using a targeted antibody array of about 30 proteins of inflammatory and neurodegenerative origin (affected voxels vs mean fluorescent intensities (MFI)).
Structural outcome vs proteomic markers in cerebrospinal fluid | Assessed at the chronic time-point (10-15 years after injury).
  Alterations at axonal and myelin integrity as assessed by magnetic resonance imaging will be associated with a proteomic profiling of cerebrospinal fluid using a targeted antibody array of about 30 proteins of inflammatory and neurodegenerative origin (affected voxels vs mean fluorescent intensities (MFI)).
Structural outcome vs auto-antibodies in serum | Assessed at the chronic time-point (10-15 years after injury).
  Alterations at axonal and myelin integrity as assessed by magnetic resonance imaging will be associated with a panel of auto-antibodies targeting central nervous system antigens ((affected voxels vs antibody titers)

SECONDARY OUTCOMES:
Acute vs chronic comparisons of proteomic markers in serum | From samples acquired in the acute phase (first weeks after injury) with samples acquired in the chronic phase (10-15 years after injury)
  Proteomic profiling using a targeted antibody array of about 30 proteins of inflammatory and neurodegenerative origin will be compared in a subset of patients between the acute and chronic stage comparing mean flourescent intensities (MFI).
Acute vs chronic comparisons of proteomic markers in CSF | From samples acquired in the acute phase (first weeks after injury) with samples acquired in the chronic phase (10-15 years after injury)
  Proteomic profiling using a targeted antibody array of about 30 proteins of inflammatory and neurodegenerative origin in CSF will be compared in a subset of patients between the acute and chronic stage comparing mean flourescent intensities (MFI).
Acute vs chronic comparisons of autoantibodies | From samples acquired in the acute phase (first weeks after injury) with samples acquired in the chronic phase (10-15 years after injury)
  A panel of auto-antibodies targeting central nervous system antigens will be compared between the acute and chronic phase (comparison of antibody titers)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to local laws and regulations, we will not be able to share IPD.